CLINICAL TRIAL: NCT00205660
Title: Changes in Adiposity and Metabolic Measures During Medication Switches to Aripiprazole From Other Atypical Antipsychotics
Brief Title: Changes in Adiposity, Metabolic Measures From Atypicals to Aripiprazole
Acronym: BMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMS #942370
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-07

CONDITIONS: Schizophrenia; Type 2 Diabetes Mellitus
Keywords: Schizophrenia; Obesity; Hyperglycemia; Dyslipidemia; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus, Type 2; Obesity; Hyperglycemia; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stayers (Other): Subjects are randomized to stay on their current antipsychotic.
  Interventions: Other: Stayers
- Switchers (Other): Subjects are randomized to switch to aripiprazole from their current antipsychotic.
  Interventions: Other: Switchers

INTERVENTIONS:
Other: Stayers — Participants remain on their current antipsychotic.
  Arms: Stayers
Other: Switchers — Subjects are randomized to switch to aripiprazole from their current antipsychotic.
  Arms: Switchers

SUMMARY:
This proposal aims to use well-validated methodologies such as dual energy x-ray absorptiometry (DEXA), frequently sampled oral glucose tolerance tests (fsOGTTs), and hyperinsulinemic euglycemic clamps to characterize the metabolic effects of 12 weeks of aripiprazole treatment following chronic pretreatment with olanzapine, quetiapine, risperidone or ziprasidone.

We hypothesize that switching to aripiprazole treatment will induce improvements in total body adiposity, inflammation (e.g., high sensitivity C-reactive protein [hsCRP]), glucose metabolism (e.g., insulin sensitivity) and lipid metabolism (e.g., fasting plasma triglyceride), in comparison to chronic pretreatment with olanzapine, risperidone and quetiapine.

DETAILED DESCRIPTION:
Schizophrenia is associated with increased rates of obesity, hyperglycemia, dyslipidemia and type 2 diabetes mellitus (T2DM), causing increased morbidity and mortality due to acute (e.g., diabetic ketoacidosis) and long-term (e.g., vascular disease) complications.1-5As a result, cardiovascular (CV) mortality remains one of the leading causes of excess mortality in patients with psychotic disorders.6,7 T2DM is characterized by disturbances in insulin secretion and insulin action at skeletal muscle (i.e., decreased glucose disposal), liver (i.e., increased glucose production) and adipose tissue (i.e., increased lipolysis), leading to disturbances in glucose and lipid metabolism. The metabolic syndrome of insulin resistance, hyperinsulinemia, dyslipidemia and abdominal adiposity usually includes a procoagulant state and endothelial dysfunction, and is strongly associated with increased CV morbidity and mortality.

Hyperglycemia was first noted in patients with schizophrenia prior to the introduction of antipsychotic medications, but glucoregulatory defects, dyslipidemia and increased adiposity are all additionally associated with both older and newer antipsychotic treatments.1 In most patients, these metabolic derangements are primarily related to increases in adiposity, although treatment effects independent of adiposity may also play a role in up to 25% of cases of new onset T2DM during antipsychotic treatment.8,9 Increased adiposity, especially visceral abdominal adiposity, is associated with insulin resistance, elevated plasma lipids, and increases in inflammatory markers. All of these conditions contribute to elevated mortality and all can be directly measured in patients treated with different medications.

Direct measures of adiposity, insulin action and secretion, plasma lipid levels and inflammation are available and have been well validated as predictors of CV disease and T2DM complications. Unfortunately, to date, studies using large population-based samples of patients taking antipsychotic medications have only used insensitive measures, like random glucose, or surrogate measures such as prescription of an oral hypoglycemic agent, to estimate the prevalence of T2DM during antipsychotic treatment. No data are available concerning insulin sensitivity and secretion, plasma lipids or inflammatory markers from large population-based samples of individuals treated with antipsychotic medications. Reviewed below, limited data are available from smaller analytic studies using sensitive measures. Despite convergent evidence for the contribution of adiposity to the metabolic derangements associated with antipsychotic treatment, investigators have only begun to use direct measures of adiposity to characterize the weight gain associated with antipsychotic treatment.

This proposal aims to use well-validated methodologies such as dual energy x-ray absorptiometry (DEXA), frequently sampled oral glucose tolerance tests (fsOGTTs), and hyperinsulinemic euglycemic clamps to characterize the metabolic effects of 12 weeks of aripiprazole treatment following chronic pretreatment with olanzapine, quetiapine, risperidone or ziprasidone.

We hypothesize that switching to aripiprazole treatment will induce improvements in total body adiposity, inflammation (e.g., high sensitivity C-reactive protein [hsCRP]), glucose metabolism (e.g., insulin sensitivity) and lipid metabolism (e.g., fasting plasma triglyceride), in comparison to chronic pretreatment with olanzapine, risperidone and quetiapine.

Aim 1: To characterize the glucoregulatory effects of 12 weeks of aripiprazole treatment.

This study hypothesizes that switching to aripiprazole treatment will be associated with statistically significant improvements in glucose metabolism (e.g., insulin sensitivity) in comparison to chronic pretreatment with olanzapine. Given the planned sample size and study duration, we hypothesize that aripiprazole treatment will be associated with numerical, but not statistically significant, improvements in comparison to pretreatment with risperidone or quetiapine. We hypothesize that aripiprazole treatment will be associated with no significant change in comparison to pretreatment with ziprasidone. These hypotheses will be evaluated by measuring insulin sensitivity and other indices via fsOGTTs and hyperinsulinemic euglycemic clamps.

Aim 2: To evaluate medication-related measures of abdominal fat, total body fat and total fat-free mass.

This study hypothesizes that switching to aripiprazole treatment will be associated with reductions in adipose tissue mass in comparison to olanzapine. We hypothesize that aripiprazole treatment will be associated with numerical, but not statistically significant, reductions in comparison to pretreatment with risperidone or quetiapine. We hypothesize that aripiprazole treatment will be associated with no change in comparison to pretreatment with ziprasidone. These hypotheses will be evaluated by measuring body composition using dual energy x-ray absorptiometry (DEXA) and anthropomorphic measurements to provide estimates of total body fat, abdominal fat and fat-free mass.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets DSM-IV criteria for Schizophrenia
* 18-60 years of age or older
* Able to give informed consent
* Treated with olanzapine, quetiapine, risperidone or ziprasidone for greater than or equal to 3 months prior to enrollment

Exclusion Criteria:

* pregnant or breastfeeding women will be excluded
* Meets DSM-IV criteria for substance abuse or dependence within past 6 months
* involuntary legal status (as per Missouri law)
* any serious medical disorder that may confound assessment of symptoms
* subjects taking prescription medications except psychotropic meds
* meets DSM-IV criteria for Mental Retardation (mild or worse)
* Subjects taking tricyclic antidepressants or mood stabilizers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2005-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W. Newcomer, MD, Principal Investigator — Washington University School of Medicine and Florida Atlantic University
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haupt DW, Newcomer JW. Hyperglycemia and antipsychotic medications. J Clin Psychiatry. 2001;62 Suppl 27:15-26; discussion 40-1. PMID 11806485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from wide range of sites in the St. Louis community. Some advertising with flyers was used however the majority of the recruitment was done using community outreach, doctor-to-doctor or self-referrals, and referrals from board and care and community support programs. All recruitment materials were approved by the IRB.
Pre-assignment Details: Participants were enrolled in the study once they signed consent. After enrollment, participants were brought in for a screening visit consisting of a diagnostic interview, screening labs, a review of records and a discussion with their primary psychiatrist. If the patient met all inclusion criteria after screening, study visits were scheduled.
Groups:
- Stayers: Participants in this arm were randomized to stay on their current antipsychotic.
- Switchers: Participants in this arm were randomized to switch to aripiprazole from their current antipsychotic.
Period: Overall Study
Arm/Group | Stayers | Switchers
Started | 14 | 37
Completed | 12 | 35
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Stay: Subjects in this group stayed on their current antipsychotic.
- Switch: Subjects in this group switched to aripiprazole from their current antipsychotic.
- Total: Total of all reporting groups
Arm/Group | Stay | Switch | Total
Number analyzed (Participants) | 14 | 37 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (7.3) | 37.4 (11.1) | 38.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 10 | 30 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 10 | 14
  Non-White | 10 | 27 | 37
Weight [Mean (Standard Deviation); unit: kilograms] | 93.7 (18.7) | 91.4 (20.1) | 92.0 (19.5)
BMI [Mean (Standard Deviation); unit: kilograms per squared meters] | 30.7 (6.7) | 30.6 (6.2) | 30.7 (6.3)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] — Population: 1 participant was missing a waist measurement.
  centimeters
    number analyzed (Participants) | 13 | 37 | 50
    (all) | 101.8 (14.0) | 103.7 (15.8) | 103.2 (15.2)
DEXA Total Fat [Mean (Standard Deviation); unit: kilograms] — Population: 1 participant was missing a DEXA.
  kilograms
    number analyzed (Participants) | 14 | 36 | 50
    (all) | 29.7 (12.5) | 26.9 (10.9) | 27.7 (11.3)
Whole Body Sensitivity [Mean (Standard Deviation); unit: mg/kg/min] | 5.8 (2.9) | 4.6 (2.7) | 4.9 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Body Fat (kg).
Description: This study hypothesizes that switching to aripiprazole treatment will be associated with reductions in adipose tissue mass in comparison to olanzapine.
Time Frame: 12 Weeks
Population: The analysis was "per protocol" and included subjects that completed both a baseline and endpoint assessment, which in this case, was a DEXA scan.
Measure: Mean (Standard Deviation); unit: change in kilograms
Groups:
- Stayers: The subjects in this arm stayed on their current antipsychotic following entry into the study.
- Switchers: The subjects in this arm switched to aripiprazole from their current antipsychotic following entry into the study.
- Total: This arm consists of pooled treatment groups (i.e., those who stayed on their current antipsychotic and those who switched to aripiprazole).
Arm/Group | Stayers | Switchers | Total
Number analyzed (Participants) | 12 | 34 | 46
change in kilograms | 0.15 (1.96) | -1.77 (2.66) | -1.27 (2.62)
Statistical Analysis 1: Comparison: Stayers vs Switchers; A repeated measures ANCOVA was used to test for a time by treatment condition interaction that would indicate differences between groups in change over time in the primary outcome. The null hypothesis was that there were no differences between groups in the change over time (time x treatment condition); Test type: Superiority; p = 0.03, ANCOVA — The a priori threshold for statistical significance in this planned primary test was p<0.05

2. Primary Outcome: Change in Whole Body Sensitivity (mg/kg/Min)
Description: This study hypothesized that switching to aripiprazole treatment will be associated with statistically significant improvements in whole body sensitivity (mg/kg/min) in comparison to chronic pretreatment with olanzapine.
Time Frame: 12 Weeks
Population: The analysis was "per protocol" and included subjects that completed both a baseline and endpoint assessment, which in this case, was a hyperinsulinemic euglycemic clamp.
Measure: Mean (Standard Deviation); unit: change in mg/kg/min
Arm/Group | Stayers | Switchers | Total
Number analyzed (Participants) | 12 | 34 | 46
change in mg/kg/min | -0.67 (1.12) | 1.19 (2.09) | 0.70 (2.05)
Statistical Analysis 1: Comparison: Stayers vs Switchers; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.01, ANCOVA — The a priori threshold for statistical significance in this planned primary test was p<0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the entire course of the 12-week study.
Groups:
- Stay: Includes subjects who stayed on their current antipsychotic throughout the study
- Switch: Includes subjects who switched to aripiprazole
Arm/Group | Stay | Switch
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/35
Other Adverse Events (participants affected / at risk) | 2/12 | 17/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stay (N=12) | Switch (N=35)
Hunger (General disorders) | 1 | 9
Drowsiness/Somnolence (General disorders) | 1 | 7
Tiredness/Fatigue (General disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No